CLINICAL TRIAL: NCT05310188
Title: Diagnostic and Prognostic Values of Cholinesterase, Amylase, Lipase and Neutrophil-to-lymphocyte Ratio in Acute Pesticide Poisoning Cases
Brief Title: Cholinesterase, Amylase, Lipase and Neutrophil-to-lymphocyte Ratio in Acute Pesticide Poisoning Cases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa AbouBakr Ahmed, director, Assiut University
Other Study IDs: Acute pesticide poisoning
Record Dates: First submitted 2022-03-01; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Pesticide Poisoning
Keywords: cholinesterease; lipase; amylase; NL ratio

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples and serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: pseudocholinesterease — blood samples
  Other Names: lipase; NLR; amylase

SUMMARY:
To estimate diagnostic levels of amylase, lipase, pseudocholinestrase and neutrophili lymphocytic ratio to different pesticide poisoning.

In addition to detect prognostic values of theses enzymes & NLR and its relation to the outcome of all pesticide poisoning.

To assess descriptive sociodemographic criteria of these poisoned cases, mode of toxicity, type of pesticide poisoning at emergency room, any other associated toxicity as well as the clinical outcome.

DETAILED DESCRIPTION:
Acute pesticide poisoning is a global health problem responsible for majority of deaths in poisoning cases.

There is a study estimated that about 385 million cases of unintentional acute pesticide poisoning occur annually world-wide including about 11,000 fatalities.

Thirty percent of global suicides are due to pesticide poisoning as they are of low cost and easily accessible.

Most common suicidal pesticide are classified according to WHO to organophosphorus insecticides, carbamate insecticide, and methyl parathion /or the herbicide paraquat.

. Aluminum phosphide(ALP) becomes one of the commonest causes of poisoning. It is extremely toxic after self-poisoning, with a case fatality often exceeding 70% after ingestion.

Severe poisoning also has the potential to induce multi-organ failure. The exact site or mechanism of its action has not been proved in humans. Rather than targeting a single organ to cause gross damage.

organophosphorus pesticides inhibit acetylcholine esterase enzyme so that lead to accumulation of Ach and muscarinic, nicotinic and central nervous system (CNS) receptor overstimulation. The severity of acute poisoning depends on level of cholinesterase.

Detection of pseudocholinestrase is a good biomarker and the most specific lab test of acute pesticide poisoning.

There is a relative relationship between plasma cholinesterase and manifestation and final outcome so that level of PChE is a good prognostic value and could help in treatment plans.

Cholinergic stimulation of pancreas leads to hyperamylasemia so amylase could be used as a prognostic tool of acute pesticide poisoning, lipase can be helpful with amylase for early detect of pancreatitis as well as determination of severity of poisoning.

The neutrophil-to-lymphocyte ratio (NLR) is an independent predictor of short- and long-term mortality in critically ill patients, and measurement is simple, cheap, and fast Furthermore, the NLR is a powerful prognostic predictor of cardiovascular affection, acute ischemic stroke, and many other diseases. So high NLR is associated with the risk of mortality of acute toxicity.

laboratory evaluation through using rapid, simple, cheap tests plays an important and vital role for confirmation of poisoning, diagnosing the first acute organ damage as well as assessing the severity of poisoning.

Emergency physicians can help in improvement of these patient and reduce deaths by accurate assessment of lab markers.

ELIGIBILITY:
Inclusion Criteria:

* All ages
* Both sex
* Any possible route of exposure to pesticides

Exclusion Criteria:

* Exposure to medications or toxic chemicals other than pesticides.
* Patients with chronic comorbidities, including liver cirrhosis, symptomatic heart failure, end stage CKD(on regular hemodialysis) and COPD.
* Patients with gallstone history or DM
* Recent abdominal trauma
* Open abdominal surgery within one year ago

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Sociodemographic criteria: age, gender, residence, occupation, level of education,
  * Toxicity associated data: mode of exposure, time of exposure, symptoms appear, any measures done to reduce the toxicity before reaching the hospital
  * Medical history (HR, BP, kidney function, liver function and blood glucose level)
  * Clinical lab result of pseudocholinesterase, amylase, lipase and neutrophil-to-lymphocyte ratio at three times.
    * the first with 6 hrs. of admission
    * the second after 24 hrs. of the treatment regimen taken
    * the third after 48 hrs
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic and prognostic values of cholinesterase in acute pesticide poisoning cases | baseline
  clinical lab result of pseudocholinesterase
diagnostic and prognostic value of amylase in acute pesticide poisoning cases | baseline
  blood level of amylase
diagnostic and prognostic value of lipase in acute pesticide poisoning cases | baseline
  blood level of lipase
diagnostic and prognostic value of neutrophil-to-lymphocyte ratio in acute pesticide poisoning case | baseline
  blood level of neutrophil-to-lymphocyte ratio

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Mohammed Abd EL-Rahman, Ass.Prof, Study Director — Assiut University; Hanan Sharaf El_Deen Mohammed, Ass.prof, Study Director — Assiut University

REFERENCES:
- [Background] Afzali S, Taheri SK, Seifrabiei M. Butyrylcholinesterase level in poisoned patients with phosphide compounds. Caspian J Intern Med. 2019 Fall;10(4):458-462. doi: 10.22088/cjim.10.4.458. PMID 31814946
- [Background] Boedeker W, Watts M, Clausing P, Marquez E. The global distribution of acute unintentional pesticide poisoning: estimations based on a systematic review. BMC Public Health. 2020 Dec 7;20(1):1875. doi: 10.1186/s12889-020-09939-0. PMID 33287770
- [Background] Mu Y, Hu B, Gao N, Pang L. Prognostic value of the neutrophil-to-lymphocyte ratio in acute organophosphorus pesticide poisoning. Open Life Sci. 2021 Jul 15;16(1):703-710. doi: 10.1515/biol-2021-0069. eCollection 2021. PMID 34307885
- [Background] Mehrpour O, Jafarzadeh M, Abdollahi M. A systematic review of aluminium phosphide poisoning. Arh Hig Rada Toksikol. 2012 Mar;63(1):61-73. doi: 10.2478/10004-1254-63-2012-2182. PMID 22450207
- [Background] Dungdung A, Kumar A, Kumar B, Preetam M, Tara RK, Saba MK. Correlation and prognostic significance of serum amylase, serum lipase, and plasma cholinesterase in acute organophosphorus poisoning. J Family Med Prim Care. 2020 Apr 30;9(4):1873-1877. doi: 10.4103/jfmpc.jfmpc_205_20. eCollection 2020 Apr. PMID 32670933